CLINICAL TRIAL: NCT00759460
Title: An Exploratory Study Conducted as an add-on to Clinical Trial 11286, to Evaluate the Metabolic Effect of up to 12 Weeks Treatment With Sertindole and Olanzapine in Patients With Schizophrenia
Brief Title: Study on Metabolic Parameters of Sertindole in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11286C
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sertindole
- 2 (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Sertindole — 12 to 20 mg daily after initial up-titration, encapsulated tablets, orally, 84 days
  Arms: 1
Drug: Olanzapine — 10 to 20 mg daily after initial up-titration, encapsulated tablets, orally, 84 days
  Other Names: Zyprexa
  Arms: 2

SUMMARY:
The purpose of this exploratory study is to evaluate the effects of sertindole and olanzapine on metabolic parameters and syndrome in patients with schizophrenia.

DETAILED DESCRIPTION:
The prevalence of metabolic syndrome is estimated to be around 20-25% of the population and is particularly high in patients with schizophrenia. Individuals with metabolic syndrome are twice as likely to die from, and three times as likely to suffer from a heart attack or stroke compared to individuals without the syndrome.

Patients on atypical antipsychotic medication should be considered a high risk group for diabetes and cardiovascular disease. Weight gain is common in patients taking neuroleptics and atypical antipsychotics, and excessive body weight is a risk factor for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia
* Participation in 11286 study
* Capable of completing all study-related activities for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline by treatment and between treatments for each of the components of the metabolic syndrome | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CN002, Beijing, China